CLINICAL TRIAL: NCT01287767
Title: A Support Program for Carers of Persons With Dementia - a 24 Months RCT
Brief Title: A Support Program for Carers of Persons With Dementia
Acronym: DIF2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Centre for Ageing and Health (Other)
Collaborators: The Research Council of Norway (Other); Kavli Research Center for Ageing and Dementia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FI09; NFR189449 (Other: The Research Counsil of Norway)
Record Dates: First submitted 2011-01-26; First posted 2011-02-01 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Dementia; Depression
Keywords: Dementia; Depression; Burden of care; Psychosocial intervention; Family home care
MeSH Terms: conditions — Dementia; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group, ordinary support (No Intervention): Home care as usual.
- A multidimensjonalt support program (Experimental): •Behavioral (e.g., Psychotherapy, Lifestyle Counseling) The family will receive individual consulting, teaching and problem solving in support groups.
  Interventions: Behavioral: A multidimensional support program

INTERVENTIONS:
Behavioral: A multidimensional support program — Counseling, education and problem-solving in support group, ad hoc counseling
  Arms: A multidimensjonalt support program

SUMMARY:
Dementia is one of the most common and devastating diseases in the elderly, it leads to helplessness, no cure exists and therefore care is necessary to provide. The care is associated with a great burden for the family carers and expensive for the society when residential care is required. The purpose of this study is to improve knowledge on how to provide better care for both the patients and their family carers, the investigators want to carry out a controlled trial using a rather cheap form of intervention, a multidimensional support program - an 18 months randomized controlled intervention study.

DETAILED DESCRIPTION:
The 230 dyads of families, patients and carers, will be recruited from 18 municipalities, 18 from each municipality with at least 15 000 inhabitants. Only home dwelling patients and carers with at least weekly face-to face contact with the patient will be included. The patients will be recruited both from memory clinics, outpatients clinics in geriatric medicine and old age psychiatry and from home nurse districts. The patients should have a diagnosis of dementia according to ICD-10 criteria, have a score on Mini Mental State Examination of at least 15 points and have capacity to give informant consent to participation in the study. The carers should score at least five on the Relatives' Stress Scale.

115 family, control group, will receive care 'as usual' in the municipalities. The 115 family intervention group will have a duration of 18 months consisting individual counselling, education about dementia, problem-solving groups and ad-hoc counselling when needed. Effects will be measured at three levels, at patient level, at carer level and at societal level. Measurements will take place at baseline, after three, six, 12 and 18 months. At patient level, the Cornell scale will be used as the primary outcome. At carer's level, the primary outcome is the Relatives' Stress Scale. For the outcome on the social level Resource Utilisation in Dementia will be used.

The carers will be contacted every year up till five years after the intervention ended to give information about their own physical and psychological health and the patient's use of formal help such as day care centre, respite care and permanent nursing home placement.

ELIGIBILITY:
Inclusion Criteria:

* Home dwelling patients and carers with at least weekly face-to face contact with the patients
* The patients should have a diagnosis of dementia according to ISD-10 criteria
* A Mini Mental State Examination (MMSE)og at least 15 point.
* Have capacity to give informant consent to participation in the study
* The carers should score at least five on the Relatives'Stress Scale(RSS)

Exclusion Criteria:

* Result from the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2009-10; Primary Completion 2013-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Differences in level of depression between groups | After 12 months
  Cornell scala for depression will be used to measure depression among the person with dementia and Geriatric Depression Scale (GDS) will be used for the carer.

SECONDARY OUTCOMES:
Resource Utilisation in Dementia | after 12 months
  Resource Utilisation in Dementia (RUD Lite) instrument (Wimo, 1998) which contains questions concerning use of community care services, type of accommodation, the employment status of the patient and primary caregiver, medical and informal care.
Change in stress among carers | after 12 months
  Relatives Stress Scale(RSS) will be used
Neuropsychiatric Inventory (NPI) | after 12 months
Quality of life among people with dementia and carers | after 12 months
  The Quality of life in Alzheimer's disease (QOL-AD)
Measures function in activities of daily living | after 12 months
  Lawton & Brody Instrumental and Performance activities daily living scale (IADL and PADL)
measure expressed emotion | after 12 months
  Using Felt Expressed Emotion Rating Scale (FEERS)
Locus of control among carers | after 12 months
Mini mental status (MMSE) | after 12 months
Differences in level of depression between groups | after 24 months
  Cornell scala for depression will be used to measure depression among the person with dementia and Geriatric Depression Scale (GDS) will be used for the carer.
Resource Utilisation in Dementia | after 24 months
Change in stress among carers(RSS) | after 24 months
Neuropsychiatric Inventory (NPI) | after 24 months
Quality of life among people with dementia and carers(QOL-AD) | after 24 months
Measures function in activities of daily living | after 24 months
Locus of control among carers | after 24 months
measure expressed emotion | after 24 months
Mini mental status (MMSE) | after 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Knut Engedal, M.D.PhD, Principal Investigator — Norwegian Centre for Ageing and Health
Locations (1):
- Norwegian Centre for Ageing and Health, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Bjorge H, Kvaal K, Ulstein I. The effect of psychosocial support on caregivers' perceived criticism and emotional over-involvement of persons with dementia: an assessor-blinded randomized controlled trial. BMC Health Serv Res. 2019 Oct 24;19(1):744. doi: 10.1186/s12913-019-4551-x. PMID 31651321